CLINICAL TRIAL: NCT04412733
Title: EFFECTIVENESS OF PULSED ULTRASOUND TREATMENT ON PATIENT WITH BELL'S PALSY, A DOUBLE-BLIND, RANDOMİZED, PLACEBO-CONTROLLED TRIAL
Brief Title: EFFECTİVENESS OF PULSED ULTRASOUND TREATMENT ON PATIENTS WITH BELL'S PALSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: meryemkaysin
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Bell Palsy
Keywords: Bell's palsy; facial paralysis; pulsed ultrasound
MeSH Terms: conditions — Bell Palsy; Facial Paralysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Ultrasound Group (Experimental): Patients in pulsed ultrasound group received pulsed ultrasound treatment (frequency: 1000 kHz, intensity: 0.5w/cm2, on-off ratio: 1:2 ) 5-min daily session, 5 days per weeks, for a total of 15 sessions.
  Interventions: Device: Therapeutic Pulsed Ultrasound
- Sham Group (Sham Comparator): Control group received sham ultrasound with the same protocol.
  Interventions: Device: Sham Ultrasound

INTERVENTIONS:
Device: Therapeutic Pulsed Ultrasound — Patients in pulsed ultrasound group received pulsed ultrasound treatment (frequency: 1000 kHz, intensity: 0.5w/cm2, on-off ratio: 1:2). Pulsed ultrasound treatment were applied with 5-cm2 head Enraf-Nonius Sonopuls 434 ultrasound device.
  Arms: Pulsed Ultrasound Group
Device: Sham Ultrasound — Control group received sham ultrasound treatment
  Arms: Sham Group

SUMMARY:
Bell's palsy (idiopathic facial palsy) is the most common peripheral lesion of the cranial nerves and the most common mono-neuropathy. Therapeutic ultrasound (US) is among the commonly used physical modalities for treating musculoskeletal disorders. The effects of US are due to alteration of cell membrane activity, vascular wall permeability and facilitation of tissue healing. The aim of this study is to investigate the effect of pulsed US treatment in patients with Bell's palsy when added to superficial heating, massage and exercise therapies.

DETAILED DESCRIPTION:
In this double -blind, randomized placebo-controlled trial, 32 patients (aged 18-65 years) diagnosed as idiopathic facial palsy with appropriate criteria were included. All patients were evaluated with motor nerve conduction studies and electromyography at 3-4 weeks after the onset of paralysis and 3 months after the treatment. Paralytic side frontalis and orbicularis oris muscles were used for electrophysiological analysis. Electrophysiological examinations were performed by an experienced electromyographer who was blind to the patient's treatments. Patients were separated into two groups as Group 1 (pulsed ultrasound therapy) and Group 2 (sham). Both groups were undergone to a conservative treatment program (20 min hot pack, massage 20 min and facial expression exercises) for 3 weeks, 5 days a week. In group 1 pulsed US treatment (frequency: 1000 kHz, intensity: 0.5w/cm2, on-off ratio: 1:2, duration 5 min) were applied to the paralyzed facial muscles. The patients in group 2 received exactly the same procedure as the treatment group, except that the power switch was off. All treatments were applied for 5 days a week for 3 weeks by the same 5-cm2 head US device (Enraf-Nonius Sonopuls 434) and the same physiotherapist. Patients were assessed at baseline, after last session, and 3 months after the treatment. Sunnybrook Facial Grading System, House Brackmann Facial Grading System and Facial Disability Index and electrophysiologic parameters were used for outcome evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Clinically diagnosed as Bell's palsy by an ear nose and throat specialist.

Exclusion Criteria:

* Central nervous system pathology
* Recurrent Bell's palsy
* Diabetes mellitus
* Contraindications of ultrasound treatment

  * Active infection
  * Cancer
  * Pregnancy
  * Lactation
  * Open wound around application area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Sunnybrook Facial Grading System | 3 months
  Sunnybrook Facial Grading System is a scale used to assess facial function, and scores range from 0 (complete paralysis) to 100 (normal facial function). This scale provides a clinical score which combines a static and dynamic assessment of facial muscles with the degree of synkinesis.
Hause Brackman Facial Nerve Grading System | 3 months
  Hause Brackman Facial Nerve Grading System is based on a six-grade score ( I-VI) that offers a gross evaluation of facial motor function and also includes evaluation of sequelae.
Facial Disability Index | 3 months
  Facial Disability Index evaluates the disability of individuals with Bell's Palsy by a total of 10 questions which assess physical and social limitations.

SECONDARY OUTCOMES:
Electrophysiologic Changes | 3 months
  Secondary outcome measures were changes of facial nerve latencies and amplitudes of compound muscle action potentials derived from the frontalis and orbicularis oris muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Yilmaz Kaysin, MD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patients were separated into two groups as Group 1 (pulsed ultrasound therapy) and Group 2 (sham). Both groups were undergone to a conservative treatment program (20 min hot pack, massage 20 min and facial expression exercises) for 3 weeks, 5 days a week. In group 1 pulsed US treatment (frequency: 1000 kHz, intensity: 0.5w/cm2, on-off ratio: 1:2, duration 5 min) were applied to the paralyzed facial muscles. The patients in group 2 received exactly the same procedure as the treatment group, except that the power switch was off. All treatments were applied for 5 days a week for 3 weeks by the same 5-cm2 head US device (Enraf-Nonius Sonopuls 434) and the same physiotherapist. Patients were assessed at baseline, after last session, and 3 months after the treatment. Sunnybrook Facial Grading System, House Brackmann Facial Grading System and Facial Disability Index and electrophysiologic parameters were used for outcome evaluation.